CLINICAL TRIAL: NCT01449994
Title: Efficacy of Instrumental Chiropractic Treatment Using Activator Methods for Pain and Dysfunction.A Randomized Placebo-controlled Clinical Study on Juvenile Athletes With Leg Pain
Brief Title: Efficacy of Instrumental Chiropractic Treatment Using Activator Methods for Pain and Dysfunction in Juvenile Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Frank Schneider, MD, senior orthopedic surgeon, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Activator in Austria
Record Dates: First submitted 2011-07-20; First posted 2011-10-10 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Pain in Leg, Unspecified; Knee Sprain
Keywords: knee; hip; ankle; foot; pain; lower limb; activator; instrumental; chiropractic; Painful functional conditions of the lower extremity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo-Activator (Placebo Comparator): Treatment with Placebo Activator IV
  Interventions: Device: Activator IV (Activator Methods Int. Phoenix, Arizona)
- Activator (Active Comparator): Treatment with Activator IV adjusting instrument
  Interventions: Device: Activator IV (Activator Methods Int. Phoenix, Arizona)

INTERVENTIONS:
Device: Activator IV (Activator Methods Int. Phoenix, Arizona) — Instruments gives a defined impulse on specified areas of the body
  Other Names: Chiropractic adjusting instrument

SUMMARY:
The goal of the study is to prove efficacy of instrumental chiropractic treatment for leg pain in juvenile athletes.

A randomized placebo controlled clinical trial including juvenile athletes with functional impairment and pain in thigh, leg or foot is performed.

Hypothesis: Instrumental chiropractic treatment with the "activator instrument "following the "activator methods" diagnostic evaluation should lead to significant improvement of complaints and functional impairment compared to the control group treated by a deactivated instrument following a sham evaluation protocol.

DETAILED DESCRIPTION:
Pain and functional impairment may force young athletes to interrupt training plans and/or even stay away from competition. Usually elite athletes run through an abundance of tests and diagnostic features-too often these high cost diagnostics don´t provide useful information for treatment. Treating the symptoms in the first place (after ruling out severe pathology) will reduce the need for extensive diagnostic routines and bring athletes back to competition earlier.

In our outpatient department of young elite sportsmen chiropractic instrumental treatment is performed routinely- mostly a pain reduction of 3-4 levels in VAS is achieved within the first session of treatment.

The following study is thought to prove the efficacy of the Chiropractic Instrumental Treatment performed at our sports-medicine outpatient department.

ELIGIBILITY:
Inclusion Criteria:

* functional problems in the lower extremities

Exclusion Criteria:

* severe pathology that requires different treatment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction of Pain | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Schneider, MD, Principal Investigator — Meical University Graz Department of pediatric orthopedics
Locations (1):
- MedUni Graz Pediatric Surgery and Ped. Orthopedics, Graz, Styria, Austria